CLINICAL TRIAL: NCT05528926
Title: Parent Training for the Treatment of Irritability in Children and Adolescents: a Multisite Randomized Controlled, 3-parallel-group, Evaluator-blinded, Superiority Trial
Brief Title: RESist Against Irritability Superiority Trial
Acronym: RESIST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RECHMPL20_0038
Record Dates: First submitted 2022-08-31; First posted 2022-09-06 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Irritable Mood
Keywords: Irritability; Parent Management Training (PMT); Non-Violent Resistance (NVR)
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: 3 parallel groups to compare:
  * Non-Violent Resistance parent training (NVR)
  * Parent Management Training (PMT)
  * Treatment As Usual (TAU)
Who Masked: Outcomes Assessor
Masking Description: In the RESIST trial, independent evaluators will be blinded to the type of program received by the parents; this aspect will be monitored throughout the study and parents will be instructed before every assessment to avoid disclosing the type of therapy received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-Violent Resistance (NVR) program (Other): The Non-Violent Resistance (NVR) parent group-format program has been designed to develop a positive form of authority based on parental presence, a parental support network, strategies of nonviolent responses which avoid escalation and reconciliation gestures.
  Interventions: Other: Non-Violent Resistance
- Parent Management Training (PMT) program based on Barkley's program for defiant children (Other): The Parent Management Treatment (PMT) program is an evidence-based treatment for disruptive behaviour disorder in which the child's social environment is modified according to principles of operant conditioning and contingency management. The parental response to the child's behaviour increases or decreases the likelihood of targeted behaviour.
  Interventions: Other: Parent Management Training
- Treatment as usual (TAU) (Other): The TAU group receives non-pharmacological and pharmacological therapies as usually provided in the participating centres but without having had a structured parent program.
  Interventions: Drug: Treatment As Usual

INTERVENTIONS:
Other: Non-Violent Resistance — The program's core features are parental self-control and emotional support. In the NVR program, parents recruit supporters to help them deal with their children's problematic behaviours. Developing emotional control means that the parent opposes non-violent resistance to his child's behaviour, not escalating the explosive situation.
  10 sessions (5 sessions per day for 2 consecutive days and two booster sessions at M1 and M3 after completion).
  Other Names: NVR program
  Arms: Non-Violent Resistance (NVR) program
Other: Parent Management Training — The gold-standard treatment for disruptive behaviour disorder in children and adolescents. The objective is to train parents to cope with the difficult situations they encounter, to teach them effective control strategies that are coherent and adapted to the 'deviant' behaviour of their children to reduce the intensity of events and their repercussions within the family.
  10 sessions (5 sessions per day for 2 consecutive days and two booster sessions at M1 and M3 after completion).
  Other Names: PMT program
  Arms: Parent Management Training (PMT) program based on Barkley's program for defiant children
Drug: Treatment As Usual — The TAU group receives non-pharmacological and pharmacological therapies as usually provided in the participating centres but without having had a structured parent program in the last 6 months assessed at baseline, M1 and M3.
  Other Names: TAU
  Arms: Treatment as usual (TAU)

SUMMARY:
Irritability is defined as developmentally inappropriate proneness to anger. Irritability is a symptom of several mental health conditions in children and adolescents such as attention deficit hyperactivity disorder (ADHD), oppositional defiant disorder (ODD), conduct disorder (CD), depressive disorders, anxiety disorders.Irritability has been associated with poor functional outcomes across the lifespan and was found to be specifically associated with concurrent and longitudinal emotional disorders, suicidality and impaired academic and socio-professional functioning. Children with high irritability also have distinct physiological profiles with hyper-reactivity to stress and perceived threats.

Despite the high prevalence and health issues related to irritability, there is little treatment research on this topic. Developing evidence-based non-pharmacological treatment options for children suffering from severe, chronic irritability is therefore a particularly important target for clinical research.

DETAILED DESCRIPTION:
Irritability is defined as developmentally inappropriate proneness to anger. Irritability is a symptom of several mental health conditions in children and adolescents such as attention deficit hyperactivity disorder (ADHD), oppositional defiant disorder (ODD), conduct disorder (CD), depressive disorders, anxiety disorders. Both tonic (e.g. negative quality of mood) and phasic (e.g. temper outbursts) irritability are criteria of the DSM-5 Disruptive Mood Dysregulation Disorder and the World Health Organization has considered the addition of a specifier to indicate whether ODD presents with chronic irritability and anger in the revision of the International Classification of Disease.

Irritability has been associated with poor functional outcomes across the lifespan and was found to be specifically associated with concurrent and longitudinal emotional disorders, suicidality and impaired academic and socio-professional functioning. Children with high irritability also have distinct physiological profiles with hyper-reactivity to stress and perceived threats.

Irritability is included in the negative valence system of RDoC as "frustrative non-reward". According to this neuroscience-based classification, irritability is an excessive response of an individual faced with the impossibility to achieve an expected goal and has been linked to dysregulations of the autonomic nervous system and the reward network. Another pathophysiological line of research conceptualizes irritability as an aberrant response to threat (e.g. irritable individuals may attack more rapidly and in broader contexts).

Despite the high prevalence and health issues related to irritability, there is little treatment research on this topic. Developing evidence-based non-pharmacological treatment options for children suffering from severe, chronic irritability is therefore a particularly important target for clinical research. One of the first steps in achieving this goal includes testing new therapies against extant interventions. Parent training programs decrease aggressive behaviours in children and are therefore good candidates for the improvement of irritability. Low parental warmth, lack of positive parental emotion socialization and high parental Expressed Emotions have been linked with irritability in children and could therefore be targeted in parental programs.

Research on the biological and psychological mechanisms mediating irritability is also needed to further improve specificity of therapeutic actions.

The project includes two ancyllary studies : RESIST-EXP and RESIST-QUAL.

* RESIST-EXP: Investigate improvement of irritability in both programs throughout emotional testing while collecting ANS functioning measurements.
* RESIST-QUAL: A qualitative interview planned after treatment completion with parents from both parent programme groups.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subject between 6 and 15 years-old.
* Express informed consent f by at least one of the parents or legal representative, and oral consent of the child.
* A confirmed K-SADS DSM-5 diagnosis of ADHD, ODD, CD, mood/anxiety disorder or DMDD, or a clinical diagnosis of IED. The request of a concomitant mental disorder allows to restrict this intervention to a clinical population.
* A Parental-rated ARI total score of 4 or above at baseline.
* A Clinical Global Impression-Severity score (CGI-S) of 4 or above (=at least moderately ill).
* Persistence of irritability symptoms 6 month or above at baseline (this avoids including children with transitory irritability).
* stable treatment regimen (pharmacological and non-pharmacological) for 2 weeks prior to inclusion and during the trial
* RESIST-QUAL : Same inclusion criteria as above with specific informed consent form signed by the participating parent.

Exclusion Criteria:

* Unavailability of parents or legal representative during the study period.
* Subjects with a DSM-5 diagnosis (clinical presentation or history) that is consistent with Schizophrenia or psychotic disorders or acute manic episodes.
* Diagnosis of Autism Spectrum Disorder (ASD) in patients who are non-verbal and with IQ lower than 70.
* Known or estimated IQ<70 or clinical diagnosis of intellectual disability.
* Subjects with severe irritability that are better accounted for by another factor, e.g.: general medical condition(s) or direct effect of a substance (i.e., medication, illicit drug use), as determined by the clinical judgment of the investigator, or related to child abuse and/or neglect.
* absence of informed consent give by at least one of the parents or legal representatives, and oral consent of the child
* inability to speak and comprehend French
* deemed unable to comply with the trial protocol
* participation in a structured parent program during the last 6 months

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 270 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline level that measure pleasure and arousal | After 3 months follow-up
  Change from baseline at 3 months after completion of the program of the Clinician-rated Affective Rating Scale (CL-ARI) assessed by blinded evaluators.
  This scale gives a range of possible scores from 0 to 12, with frequency and duration of temper outbursts quantified across three different levels of severity: mild, moderate and severe the higher the score.

SECONDARY OUTCOMES:
Secondary efficacy endpoint at 1-month follow-up | After 1 month follow-up
  Change from baseline at 1 month after completion of the program of the Clinician-rated Affective Rating Scale (CL-ARI) by blinded evaluators.
  This scale gives a range of possible scores from 0 to 12, with frequency and duration of temper outbursts quantified across three different levels of severity: mild, moderate and severe the higher the score.
Secondary efficacy endpoints at 1 and 3-month follow-up | Between 1 and 3-month follow-up
  Clinical Global Impression Improvement (CGI-I) scale from 1 to 7. the CGI-I 7-point scale to rate the patients' total improvement based on comparison with their baseline assessment from 1 = very much improved to 7 = very much worse.
Secondary efficacy endpoints at 1 and 3-month follow-up | Between 1 and 3-month follow-up
  Change from baseline in the Parenting and Familial Adjustement Scale (PAFAS)
Secondary efficacy endpoints at 1 and 3-month follow-up | Between 1 and 3-month follow-up
  Change from baseline in Parent-rated ARI and Child-rated Cranky thermometers
Exploratory efficacy endpoints and putative moderators and mediators. | After 3-month follow-up
  Initial score and change from baseline in expressed emotions and reflexivity during the online five-minute speech sample (FMSS) at 3 months
Exploratory efficacy endpoints and putative moderators and mediators. | At 1 month and 3 months follow-up
  Initial score and change from baseline in The Child Behavior Checklist for Ages 6-18 (CBCL 6-18) (parent-rated)
Exploratory efficacy endpoints and putative moderators and mediators. | After 3 months follow-up
  Initial scores of personality dimensions assessed with Hierarchical Personality Inventory for Children (HiPIC)
Exploratory efficacy endpoints and putative moderating and mediating variables. | At 3 months follow-up
  Initial score and change from baseline in parental expressed emotions and reflexivity rated with the Five-Minute Speech Sample (FMSS).
  The FMSS is scored by considering the following 5 categories: initial statement, relationship, criticism, dissatisfaction and emotional overinvolvement.
  * Initial statement is scored as positive, neutral, or negative
  * Relationship is scored as positive, neutral, or negative
  * Criticism is scored by a frequency count used to score the number of criticisms present in the language sample.
  * Dissatisfaction is scored as present or absent
  * Emotional overinvolvement is based on the following 5 categories:
    * selfsacrificing overprotective behavior ,
    * emotional display ,
    * statements of attitude,
    * excessive detail and/or irrelevant information about the past,
    * excessive praise.
Endpoints of the ancillary study: RESIST-EXP | At baseline ans at 3 months follow-up
  These parameters will be measured on a sub-group of patients by a wristband "E4 wristband" permitting real-time physiological data acquisition:
  Blood Volume Pulse (BVP) in L/min
Endpoints of the ancillary study: RESIST-EXP | At baseline ans at 3 months follow-up
  These parameters will be measured on a sub-group of patients by a wristband "E4 wristband" permitting real-time physiological data acquisition:
  Motor Activity (in steps/day)
Endpoints of the ancillary study: RESIST-EXP | At baseline ans at 3 months follow-up
  These parameters will be measured on a sub-group of patients by a wristband "E4 wristband" permitting real-time physiological data acquisition:
  Skin conductance (in Micro Siemens)
Endpoints of the ancillary study: RESIST-EXP | At baseline ans at 3 months follow-up
  These parameters will be measured on a sub-group of patients by a wristband "E4 wristband" permitting real-time physiological data acquisition:
  Skin temperature (in °C)
Endpoints of the ancillary study: RESIST-QUAL | After 3 months follow-up
  Acceptability (questionnaire for all parents and qualitative interview in a subsample

CONTACTS AND LOCATIONS:
Locations (1):
- UH of Montpellier, Montpellier, France

REFERENCES:
- [Derived] Fongaro E, Picot MC, Stringaris A, Belloc C, Verissimo AS, Franc N, Purper-Ouakil D. Parent training for the treatment of irritability in children and adolescents: a multisite randomized controlled, 3-parallel-group, evaluator-blinded, superiority trial. BMC Psychol. 2022 Nov 22;10(1):273. doi: 10.1186/s40359-022-00984-5. PMID 36414963